CLINICAL TRIAL: NCT01617434
Title: The Effect of Liraglutide Versus Placebo When Added to Basal Insulin Analogues With or Without Metformin in Subjects With Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NN2211-3917; 2011-002696-41 (EudraCT Number); U1111-1121-9874 (Other: WHO)
Record Dates: First submitted 2012-06-08; First posted 2012-06-12 (Estimated); Results first posted 2014-10-28 (Estimated); Last update posted 2017-03-08 (Actual); Status verified 2017-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Liraglutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Liraglutide (Experimental)
  Interventions: Drug: liraglutide
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: liraglutide — Maximum 1.8 mg administered s.c. (subcutaneously, under the skin) once daily in addition to the subject's stable pre-trial basal insulin analogue regimen plus/minus metformin.
  Arms: Liraglutide
Drug: placebo — Placebo administered s.c. (subcutaneously, under the skin) once daily in addition to the subject's stable pre-trial basal insulin analogue regimen plus/minus metformin.
  Arms: Placebo

SUMMARY:
This trial is conducted in Asia, Europe and North and South America. The aim of the trial is to investigate the effect of liraglutide versus placebo when added to basal insulin analogues with or without metformin in subjects with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with type 2 diabetes for at least 180 days prior to screening and treated with stable basal insulin analogue dose of minimum 20 U/day with or without stable metformin equal to or above 1500 mg/day for at least 8 weeks prior to screening (defined as insulin adjustments less than 10% during the past 8 weeks as assessed by the investigator)
* HbA1c (glycosylated haemoglobin A1c) 7.0-10.0% (both inclusive)
* Body mass index (BMI) 20-45 kg/m^2 (both inclusive)

Exclusion Criteria:

* Female of child-bearing potential who is pregnant, breast-feeding or intending to become pregnant
* Recurrent severe hypoglycaemic episodes or hypoglycaemic unawareness
* Treatment with glucose-lowering agent(s) other than stated in the inclusion criteria in a period of 12 weeks prior to screening
* Impaired liver or renal function
* Uncontrolled treated or untreated hypertension (systolic blood pressure (SBP) equal to or above 180 mmHg and/or diastolic blood pressure (DBP) equal to or above 100 mmHg)
* Any clinically significant disorder, except for conditions associated with type 2 diabetes history which in the investigator's opinion could interfere with results of the trial
* Known or suspected abuse of alcohol or narcotics

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 451 (Actual)
Dates: Start 2012-09; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (82):
- United States (30):
  - Novo Nordisk Investigational Site, Phoenix, Arizona
  - Novo Nordisk Investigational Site, Anaheim, California
  - Novo Nordisk Investigational Site, Fresno, California
  - Novo Nordisk Investigational Site, Los Angeles, California
  - Novo Nordisk Investigational Site, San Mateo, California
  - Novo Nordisk Investigational Site, San Ramon, California
  - Novo Nordisk Investigational Site, Tustin, California
  - Novo Nordisk Investigational Site, Ventura, California
  - Novo Nordisk Investigational Site, Walnut Creek, California
  - Novo Nordisk Investigational Site, Kissimmee, Florida
  - Novo Nordisk Investigational Site, Gurnee, Illinois
  - Novo Nordisk Investigational Site, Greenfield, Indiana
  - Novo Nordisk Investigational Site, Lexington, Kentucky
  - Novo Nordisk Investigational Site, Metairie, Louisiana
  - Novo Nordisk Investigational Site, Rockville, Maryland
  - Novo Nordisk Investigational Site, Methuen, Massachusetts
  - Novo Nordisk Investigational Site, Omaha, Nebraska
  - Novo Nordisk Investigational Site, Newington, New Hampshire
  - Novo Nordisk Investigational Site, Greensboro, North Carolina
  - Novo Nordisk Investigational Site, McMurray, Pennsylvania
  - Novo Nordisk Investigational Site, Spartanburg, South Carolina
  - Novo Nordisk Investigational Site, Kingsport, Tennessee
  - Novo Nordisk Investigational Site, Dallas, Texas
  - Novo Nordisk Investigational Site, San Antonio, Texas
  - Novo Nordisk Investigational Site, Sugarland, Texas
  - Novo Nordisk Investigational Site, Salt Lake City, Utah
  - Novo Nordisk Investigational Site, Midlothian, Virginia
  - Novo Nordisk Investigational Site, Richmond, Virginia
  - Novo Nordisk Investigational Site, Renton, Washington
  - Novo Nordisk Investigational Site, Martinsburg, West Virginia
- Argentina (3):
  - Novo Nordisk Investigational Site, Buenos Aires
  - Novo Nordisk Investigational Site, Caba
  - Novo Nordisk Investigational Site, Córdoba
- Canada (10):
  - Novo Nordisk Investigational Site, Coquitlam, British Columbia
  - Novo Nordisk Investigational Site, Vancouver, British Columbia
  - Novo Nordisk Investigational Site, Burlington, Ontario
  - Novo Nordisk Investigational Site, Hamilton, Ontario
  - Novo Nordisk Investigational Site, Mississauga, Ontario
  - Novo Nordisk Investigational Site, Ottawa, Ontario
  - Novo Nordisk Investigational Site, Smiths Falls, Ontario
  - Novo Nordisk Investigational Site, Thunder Bay, Ontario
  - Novo Nordisk Investigational Site, Toronto, Ontario
  - Novo Nordisk Investigational Site, Westmount, Quebec
- Finland (5):
  - Novo Nordisk Investigational Site, Helsinki
  - Novo Nordisk Investigational Site, Kerava
  - Novo Nordisk Investigational Site, Tampere
  - Novo Nordisk Investigational Site, Turku
  - Novo Nordisk Investigational Site, Ylitornio
- Germany (10):
  - Novo Nordisk Investigational Site, Aschaffenburg
  - Novo Nordisk Investigational Site, Bad Lauterberg im Harz
  - Novo Nordisk Investigational Site, Berlin
  - Novo Nordisk Investigational Site, Friedrichsthal
  - Novo Nordisk Investigational Site, Gelnhausen
  - Novo Nordisk Investigational Site, Gifhorn
  - Novo Nordisk Investigational Site, Hohenmölsen
  - Novo Nordisk Investigational Site, Mannheim
  - Novo Nordisk Investigational Site, Mayen
  - Novo Nordisk Investigational Site, Oldenburg
- India (10):
  - Novo Nordisk Investigational Site, Visakhapatnam, Andhra Pradesh
  - Novo Nordisk Investigational Site, Rohtak, Haryana
  - Novo Nordisk Investigational Site, Bangalore, Karnataka
  - Novo Nordisk Investigational Site, Indore, Madhya Pradesh
  - Novo Nordisk Investigational Site, Mumbai, Maharashtra
  - Novo Nordisk Investigational Site, Jaipur, Rajasthan
  - Novo Nordisk Investigational Site, Kolkata, West Bengal
  - Novo Nordisk Investigational Site, Hyderabad
  - Novo Nordisk Investigational Site, Kolkata
  - Novo Nordisk Investigational Site, Thriruvananthapuram
- Mexico (2):
  - Novo Nordisk Investigational Site, Pachuca, Hidalgo
  - Novo Nordisk Investigational Site, Mexico City, México, D.F.
- Netherlands (11):
  - Novo Nordisk Investigational Site, Almere Stad
  - Novo Nordisk Investigational Site, Breda
  - Novo Nordisk Investigational Site, Eindhoven
  - Novo Nordisk Investigational Site, Groningen
  - Novo Nordisk Investigational Site, Hoogeveen
  - Novo Nordisk Investigational Site, Leiden
  - Novo Nordisk Investigational Site, Rotterdam
  - Novo Nordisk Investigational Site, Velp
  - Novo Nordisk Investigational Site, Venlo
  - Novo Nordisk Investigational Site, Zoetermeer
  - Novo Nordisk Investigational Site, Zwijndrecht
- Novo Nordisk Investigational Site, Niš, Serbia

REFERENCES:
- [Result] Ahmann A, Rodbard HW, Rosenstock J, Lahtela JT, de Loredo L, Tornoe K, Boopalan A, Nauck MA; NN2211-3917 Study Group. Efficacy and safety of liraglutide versus placebo added to basal insulin analogues (with or without metformin) in patients with type 2 diabetes: a randomized, placebo-controlled trial. Diabetes Obes Metab. 2015 Nov;17(11):1056-64. doi: 10.1111/dom.12539. Epub 2015 Sep 10. PMID 26179619
- [Result] Freemantle N, Mamdani M, Vilsboll T, Kongso JH, Kvist K, Bain SC. IDegLira Versus Alternative Intensification Strategies in Patients with Type 2 Diabetes Inadequately Controlled on Basal Insulin Therapy. Diabetes Ther. 2015 Dec;6(4):573-591. doi: 10.1007/s13300-015-0142-y. Epub 2015 Nov 18. PMID 26582052
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 76 sites in 9 countries i.e. 3 sites in Argentina; 9 sites in Canada; 5 sites in Finland; 9 sites in Germany; 9 sites in India; 2 sites in Mexico; 7 sites in Netherlands; 3 sites in Serbia; 29 sites in United States.
Groups:
- Liraglutide: Liraglutide was administered subcutaneously (s.c. injection, under the skin) once daily (OD) for 26 weeks in combination with pre-trial basal insulin analogue regimen ± metformin. The starting dose of the liraglutide was 0.6 mg/day; dose was escalated to 1.2 mg/day after one week and 1.8 mg/day after 2 weeks; dose was maintained at 1.8 mg day for subsequent weeks until the end of the trial. All subjects continued their pre-trial insulin therapy of insulin glargine (100 U/mL, s.c. injection) or insulin detemir (100 U/mL, s.c. injection). Oral anti diabetic drug metformin was administered as a tablet with a total daily dose of ≥1500 mg, divided into one to three doses per day.
- Placebo: Placebo was administered subcutaneously (s.c. injection, under the skin) once daily (OD) for 26 weeks in combination with pre-trial basal insulin analogue regimen ± metformin. The starting dose of the placebo was 0.6 mg/day; dose was escalated to 1.2 mg/day after one week and 1.8 mg/day after 2 weeks; dose was maintained at 1.8 mg day for subsequent weeks until the end of the trial. All subjects continued their pre-trial insulin therapy of insulin glargine (100 U/mL, s.c. injection) or insulin detemir (100 U/mL, s.c. injection). Oral anti diabetic drug metformin was administered as a tablet with a total daily dose of ≥1500 mg, divided into one to three doses per day.
Period: Overall Study
Arm/Group | Liraglutide | Placebo
Started | 226 | 225
Exposed | 225 | 225
Completed | 191 | 174
Not Completed | 35 | 51
Not completed — Adverse Event | 12 | 3
Not completed — Protocol Violation | 8 | 7
Not completed — Withdrawal Criteria | 12 | 37
Not completed — Unclassified | 3 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Liraglutide | Placebo | Total
Number analyzed (Participants) | 225 | 225 | 450
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.3 (9.2) | 57.5 (11.1) | 58.4 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 105 | 89 | 194
  Male | 120 | 136 | 256
Body Weight [Mean (Standard Deviation); unit: kg] | 90.23 (19.98) | 91.85 (21.33) | 91.04 (20.66)
Fasting Plasma Glucose (FPG) [Mean (Standard Deviation); unit: mmol/L] | 8.32 (2.89) | 8.21 (2.90) | 8.27 (2.89)
Glycosylated Haemoglobin (HbA1c) [Mean (Standard Deviation); unit: percentage of glycosylated haemoglobin] | 8.22 (0.81) | 8.28 (0.90) | 8.25 (0.86)

OUTCOME MEASURES:

1. Primary Outcome: Change in Glycosylated Haemoglobin (HbA1c) From Baseline to Week 26
Description: The estimated mean change from baseline in HbA1c after 26 weeks of treatment.
Time Frame: Week 0 to Week 26
Population: Full analysis set (FAS) included all randomised subjects who received at least one dose of trial product (liraglutide or placebo) and who provided at least one post-baseline efficacy value. 215 subjects in the liraglutide arm and 217 subjects in the placebo arm contributed to the statistical analysis.
Measure: Mean (Standard Deviation); unit: percentage of glycosylated haemoglobin
Arm/Group | Liraglutide | Placebo
Number analyzed (Participants) | 215 | 217
percentage of glycosylated haemoglobin | -1.30 (1.015) | -0.11 (1.088)
Statistical Analysis 1: Comparison: Liraglutide vs Placebo; The null hypothesis of no difference between the two treatment arms with regard to changes from baseline in HbA1c (%) after 26 weeks of randomised treatment was analysed using a mixed model repeated measurements (MMRM) analysis with treatment, country, stratification groups as factors and baseline HbA1c as a covariate, all nested within visit; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = -1.19, 95% CI [-1.39 to -0.99]

2. Secondary Outcome: Change in Fasting Plasma Glucose (FPG) From Baseline to Week 26
Description: The estimated mean change from baseline in FPG after 26 weeks of treatment.
Time Frame: Week 0 to Week 26
Population: Full analysis set (FAS) included all randomised subjects who received at least one dose of trial product (liraglutide or placebo) and who provided at least one post-baseline efficacy value. 213 subjects in the liraglutide arm and 217 subjects in the placebo arm contributed to the statistical analysis.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Liraglutide | Placebo
Number analyzed (Participants) | 213 | 217
mmol/L | -1.44 (2.494) | -0.16 (3.006)
Statistical Analysis 1: Comparison: Liraglutide vs Placebo; The response was analysed using a mixed model repeated measurements (MMRM) analysis with treatment, country, stratification groups as factors and baseline as a covariate, all nested within visit; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = -1.28, 95% CI [-1.70 to -0.86]

3. Secondary Outcome: Change in Mean Self-Measured Plasma Glucose (SMPG) of 7-Point Profile From Baseline to Week 26
Description: The estimated mean change from baseline in mean SMPG of 7-point profile (7-points were before breakfast, 90 minutes after start of breakfast, before lunch, 90 minutes after start of lunch, before dinner, 90 minutes after start of dinner and at bedtime) after 26 weeks of treatment.
Time Frame: Week 0 to Week 26
Population: Full analysis set (FAS) included all randomised subjects who received at least one dose of trial product (liraglutide or placebo) and who provided at least one post-baseline efficacy value. 191 subjects in the liraglutide arm and 196 subjects in the placebo arm contributed to the statistical analysis.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Liraglutide | Placebo
Number analyzed (Participants) | 191 | 196
mmol/L | -2.61 (2.248) | -1.02 (3.061)
Statistical Analysis 1: Comparison: Liraglutide vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = -1.59, 95% CI [-2.01 to -1.18]

4. Secondary Outcome: Change in Body Weight From Baseline to Week 26
Description: The estimated mean change in body weight after 26 weeks of treatment.
Time Frame: Week 0 to Week 26
Population: Full analysis set (FAS) included all randomised subjects who received at least one dose of trial product (liraglutide or placebo) and who provided at least one post-baseline efficacy value. 215 subjects in the liraglutide arm and 216 subjects in the placebo arm contributed to the statistical analysis.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Liraglutide | Placebo
Number analyzed (Participants) | 215 | 216
kg | -3.54 (3.669) | -0.42 (3.909)
Statistical Analysis 1: Comparison: Liraglutide vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = -3.11, 95% CI [-3.85 to -2.37]

5. Secondary Outcome: Number of Subjects Achieving HbA1c Below 7.0% (American Diabetes Association [ADA] Target)
Description: Number of subjects achieving HbA1c below 7.0% (American Diabetes Association [ADA] target) after 26 weeks of treatment
Time Frame: At Week 26
Population: Full analysis set (FAS) included all randomised subjects who received at least one dose of trial product (liraglutide or placebo) and who provided at least one post-baseline efficacy value. 211 subjects in the liraglutide arm and 217 subjects in the placebo arm contributed to the statistical analysis.
Measure: Number; unit: percentage of subjects
Arm/Group | Liraglutide | Placebo
Number analyzed (Participants) | 211 | 217
percentage of subjects | 59.24 | 14.02
Statistical Analysis 1: Comparison: Liraglutide vs Placebo; This endpoint was analysed using a logistic regression model with treatment and stratification factors as fixed factors and the HbA1c value at baseline as a covariate. Subjects previously treated with insulin detemir without the use of metformin were not included in the analysis due to the small size of the stratum; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 8.91, 95% CI [5.45 to 14.59]

6. Secondary Outcome: Number of Subjects Achieving HbA1c Below or Equal to 6.5% (American Association of Clinical Endocrinologists [AACE] Target)
Description: Number of subjects achieving HbA1c below or equal to 6.5% (American Association of Clinical Endocrinologists [AACE] target) after 26 weeks of treatment.
Time Frame: At Week 26
Population: Full analysis set (FAS) included all randomised subjects who received at least one dose of trial product and who provided at least one post-baseline efficacy value. 211 subjects in the liraglutide arm and 217 subjects in the placebo arm contributed to the statistical analysis.
Measure: Number; unit: percentage of subjects
Arm/Group | Liraglutide | Placebo
Number analyzed (Participants) | 211 | 217
percentage of subjects | 42.91 | 3.60
Statistical Analysis 1: Comparison: Liraglutide vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 20.12, 95% CI [9.92 to 40.84]

7. Secondary Outcome: Number of Adverse Events (AEs) During The Randomised Treatment Period
Description: An AE was defined as treatment emergent if the onset date (or increase in severity) was on or after the first day of exposure to randomised treatment and no later than 7 days after the last day of randomised treatment. The adverse events were categorised as 'serious' and 'non-serious' adverse events. Adverse events were also categorised according to the severity as 'mild', 'moderate' and 'severe' adverse events.
Time Frame: Week 0 to Week 26 + 7 days follow up
Population: Safety analysis set includes all subjects who received at least one dose of the trial product.
Measure: Number; unit: Events/1000 years of patient exposure
Arm/Group | Liraglutide | Placebo
Number analyzed (Participants) | 225 | 225
Events/1000 years of patient exposure
  Adverse Events | 4918 | 3737
  Serious Adverse Events | 149 | 101
  Severe Adverse Events | 169 | 101
  Moderate Adverse Events | 1274 | 1060
  Mild Adverse Events | 3474 | 2575

8. Secondary Outcome: Number of Minor Hypoglycaemic Episodes During The Randomised Treatment Period
Description: A minor hypoglycaemic episode was defined as either, (a) an episode with symptoms consistent with hypoglycaemia with confirmation by blood glucose <2.8 mmol/L (50 mg/dL) or plasma glucose <3.1 mmol/L (56 mg/dL) that was handled by the subject him/herself or (b) any asymptomatic blood glucose value <2.8 mmol/L (50 mg/dL) or plasma glucose value <3.1 mmol/L (56 mg/dL).
Time Frame: Week 0 to Week 26 + 7 days follow up
Population: Safety analysis set includes all subjects who received at least one dose of the trial products.
Measure: Number; unit: Events/100 years of patient exposure
Arm/Group | Liraglutide | Placebo
Number analyzed (Participants) | 225 | 225
Events/100 years of patient exposure | 126 | 83

9. Secondary Outcome: Number of Severe Hypoglycaemic Episodes During The Randomised Treatment Period
Description: Severe hypoglycaemia episode was defined as an episode requiring assistance of another person to actively administer carbohydrate, glucagon or other resuscitative actions.
Time Frame: Week 0 to Week 26 + 7 days follow up
Population: Safety analysis set includes all subjects who received at least one dose of the trial products.
Measure: Number; unit: Events/100 years of patient exposure
Arm/Group | Liraglutide | Placebo
Number analyzed (Participants) | 225 | 225
Events/100 years of patient exposure | 0 | 0

ADVERSE EVENTS:
Time Frame: Week 0 to Week 26 + 7 days follow up
Description: Safety analysis set includes all subjects who received at least one dose of the trial product.
Arm/Group | Liraglutide | Placebo
Serious Adverse Events (participants affected / at risk) | 11/225 | 7/225
Other Adverse Events (participants affected / at risk) | 103/225 | 46/225
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Liraglutide (N=225) | Placebo (N=225)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 2 (2)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Arthritis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis staphylococcal (Infections and infestations) | 1 (1) | 0 (0)
Ear infection (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Genital herpes (Infections and infestations) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Incisional hernia (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Electrocardiogram change (Investigations) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Squamous cell carcinoma of the tongue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Intercostal neuralgia (Nervous system disorders) | 0 (0) | 1 (1)
Post-traumatic stress disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Percutaneous coronary intervention (Surgical and medical procedures) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Liraglutide (N=225) | Placebo (N=225)
Diarrhoea (Gastrointestinal disorders) | 24 (29) | 11 (14)
Dyspepsia (Gastrointestinal disorders) | 16 (20) | 2 (2)
Nausea (Gastrointestinal disorders) | 50 (62) | 7 (8)
Vomiting (Gastrointestinal disorders) | 20 (28) | 2 (3)
Influenza (Infections and infestations) | 8 (11) | 16 (21)
Nasopharyngitis (Infections and infestations) | 13 (19) | 14 (16)
Lipase increased (Investigations) | 16 (16) | 5 (5)
Decreased appetite (Metabolism and nutrition disorders) | 22 (22) | 5 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 12 (13) | 12 (13)
Headache (Nervous system disorders) | 8 (9) | 16 (20)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Novo Nordisk maintains the right to be informed of plans by any investigator to publish and to review any scientific paper, presentation, communication or other information concerning the investigation described in this protocol. Any such communication must be submitted in writing to the Novo Nordisk trial manager before submission for comments. Comments will be given within four weeks from receipt of the planned communication.